CLINICAL TRIAL: NCT06394050
Title: Utilizing Label-free Raman Spectroscopy for Discrimination Between Breast Cancer Tumor and Adjacent Tissues in Patients After Neoadjuvant Treatment
Brief Title: Label-free Raman Spectroscopy for Discrimination Between Breast Cancer Tumor and Adjacent Tissues After Neoadjuvant Treatment
Status: Not yet recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Jinsong Lu, Chief of Department of Breast Surgery, RenJi Hospital
Other Study IDs: KY2020-060-01
Record Dates: First submitted 2024-04-28; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Diagnosis
MeSH Terms: conditions — Disease | interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast cancer patients after neoadjuvant treatment
  Interventions: Diagnostic Test: Diagnostic Test

INTERVENTIONS:
Diagnostic Test: Diagnostic Test — there is no intervention

SUMMARY:
After neoadjuvant therapy, the primary lesion in breast cancer patients may experience tumor regression, which increases the difficulty of distinguishing between breast cancer and adjacent tissues. Raman spectroscopy is a form of scattering spectroscopy, which offers rapid and sensitive analysis, delivering detailed biochemical information and molecular signatures of internal molecular components within the sample. This study aims to discern between cancer and adjacent tissues after neoadjuvant therapy in breast cancer patients using label-free Raman spectroscopy.

ELIGIBILITY:
Inclusion Criteria:

* (1) aged ≥ 18 years; (2) histologically confirmed invasive breast cancer (clinical tumor stage T1 to T4, nodal stage N1-3, and metastasis stage M0); (3) previous treatment with neoadjuvant chemotherapy with or without target therapy (such as trastuzumab, pertuzumab), or endocrine therapy; (4) enough frozen samples of breast cancer tumor and adjacent tissue.

Exclusion Criteria:

* (1) undergoing sentinel lymph node biopsy with indocyanine green dye or methylene blue injection after neoadjuvant therapy; (2) Breast cancer during pregnancy and lactation, inflammatory breast cancer.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with local advanced breast cancer who had completed surgery after neoadjuvant therapy from Renji Hospital, School of Medicine, Shanghai Jiao Tong University.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-05-15 (Estimated); Study Completion 2024-05-20 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance | Baseline
  Area under curve, accuracy, sensitivity, specificity,

REFERENCES:
- [Background] Vanna R, Morasso C, Marcinno B, Piccotti F, Torti E, Altamura D, Albasini S, Agozzino M, Villani L, Sorrentino L, Bunk O, Leporati F, Giannini C, Corsi F. Raman Spectroscopy Reveals That Biochemical Composition of Breast Microcalcifications Correlates with Histopathologic Features. Cancer Res. 2020 Apr 15;80(8):1762-1772. doi: 10.1158/0008-5472.CAN-19-3204. Epub 2020 Feb 24. PMID 32094303